CLINICAL TRIAL: NCT00483873
Title: Phase IIB Study of Novel Quantitative Neurodiagnostic Technology in the Early Period After Cardiac Arrest
Brief Title: Cardiac Arrest Recovery EEG Study
Acronym: CARES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Infinite Biomedical Technologies (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Johns Hopkins Bloomberg School of Public Health (Other); Johns Hopkins University (Other); Medical College of Wisconsin (Other); Virginia Commonwealth University (Other)
Responsible Party: Dr. Neil Rothman, Vice-President of Research and Development, IInfinite Biomedical Technologies, llc
Other Study IDs: R44HL070129 (NIH); R44HL070129 (NIH)
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Cardiac Arrest; Arrhythmia
Keywords: Cardiac Arrest, Neurological Recovery, EEG, Quantitative EEG
MeSH Terms: conditions — Heart Arrest; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the study is to collect EEG's as close to the cardiac arrest as possible using a standard hospital EEG machine and an investigational EEG device to help determine the neurological status of the cardiac arrest patient and to help decide on possible treatment and chance of recovery. The investigational EEG machine will be simple to operate as well as easy to interpret for the clinician and the nurses. It is not to replace the electrophysiologist interpretation but to determine ealy on if further evaluation and treatment can help the patient.

DETAILED DESCRIPTION:
Cardiac arrest claims over 450,000 lives per year in the United States alone. There is a high incidence of neurological complications amongst survivors, and these represent the leading cause of morbidity.

Over the past several years, the care of these patients has been improved via the introduction of new systemic as well as neurospecific therapies. Speed of institution of therapy appears to be an important factor affecting efficacy. Yet, in the crucial initial hours to days post-arrest, assessment of neurological status in these patients is essentially non-existent.

Thus, there is a need for an objective validated tool to assess prognosis and to track neurological status in the early recovery period. In response to this need, we have developed an EEG based Cortical Health Index (CHI). This EEG-based index incorporates multiple weighted parameters derived from 2 channels (4 scalp electrodes + 1 ground electrode) which are related to neurologic functional recovery. The strength and uniqueness of this approach results from consideration of both the temporal as well as the spectral domains of EEG. Our Phase II results demonstrate that CHI measured within the first 6-hours post-arrest resuscitation is strongly correlated with clinical outcome at hospital discharge in a 30-patient cardiac arrest study. Together with our industry collaborator, we now propose to pursue regulatory approval of the CHI Monitor. Our plan involves a prospective clinical trial involving 4 centers and 100 patients (64 Cardiac Arrest Patients and 36 patients undergoing ICD placement as controls). We will test the ability of CHI to: 1) provide early prediction of subsequent neurological functional outcome of cardiac arrest patients, and 2) provide real-time tracking of brain injury and response to therapy. Successful completion of this project is defined by FDA clearance of the CHI Monitor.

It is our goal that the CHI Monitor will identify patients who could benefit from aggressive intervention, and then track the response to the therapy. Providing this information to the treating physician in the immediate post-resuscitation period represents a major change in care delivery for the cardiac arrest survivor.

ELIGIBILITY:
Inclusion Criteria:

Cardiac Arrest:

* Patients 18 years and older:

  1. with cardiac arrest in the hospital and successfully resuscitated, or
  2. with cardiac arrest out of the hospital and successfully resuscitated

ICD patients:

* Patients 18 years and older:

  1. Who are undergoing elective procedure in the electrophysiology laboratory for placement of a cardiac defibrillator and who will most likely undergo induction of ventricular arrhythmia as part of the procedure

Exclusion Criteria:

Cardiac Arrest:

1. Cardiac arrest and a known pre-existing cerebral pathology such as brain tumor, cerebral hemorrhage, encephalitis or immediately post-op neurosurgery.
2. CNS infection
3. Skull defects and scalp diseases that are not amenable to standard EEG testing

ICD patients:

1. Known pre-existing cerebral pathology such as brain tumor, cerebral hemorrhage, encephalitis or immediately post-op neurosurgery.
2. CNS infection
3. Skull defects and scalp diseases that are not amenable to standard EEG testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the hospital after out-of-hospital Cardiac arrest or for an ICD placement
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-08; Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Neil S Rothman, PhD, Principal Investigator — Infinite Biomedical Technologies - Study Sponsor; Romergryko Geocadin, MD, Principal Investigator — Johns Hopkins University; Michel Torbey, MD, MPH, Principal Investigator — Medical College of Wisconsin; Mary Ann Peberdy, MD, Principal Investigator — Virginia Commonwealth University
Locations (4):
- United States (4):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Virginia Commonwealth University, Richmond, Virginia
  - Medical College of Wisconsin at Froedtert Memorial Luthern Hospital Clinics - Neurology, Milwaukee, Wisconsin